CLINICAL TRIAL: NCT00551109
Title: A Phase II, Multi-Centre, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Safety and Efficacy of Treatment With SA4503, Once Daily for 8 Weeks, in Subjects With Major Depressive Disorder
Brief Title: SA4503 8-Week Study in Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M's Science Corporation (Industry)
Responsible Party: Kazunori Yoshikawa, M's Science Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ME1-1; EudraCT number: 2007-002740-16
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- P (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- A1 (Experimental): SA4503
  Interventions: Drug: SA4503 Low
- A2 (Experimental): SA4503
  Interventions: Drug: SA4503 High

INTERVENTIONS:
Drug: placebo — placebo, oral administration, once daily for 8 weeks
  Arms: P
Drug: SA4503 Low — Low dose, oral administration, once daily for 8 weeks
  Arms: A1
Drug: SA4503 High — High dose, oral administration, once daily for 8 weeks
  Arms: A2

SUMMARY:
The purpose of this study is to determine the efficacy of SA4503 compared to placebo in the treatment of subjects with major depressive disorder (MDD). Secondary, to evaluate the safety of SA4503 compared to placebo in subjects with MDD.

DETAILED DESCRIPTION:
Further study details as provided by M's Science Corporation:

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 65 (inclusive)
* Diagnosis of MDD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria and a shortened MINI evaluation
* HAM-D17 score of >/= 21 and a severity score of at least 2 for Item 1 (depressed mood) at both Screening and Baseline
* Current depressive episode of at least 3 months duration, and significant depressed mood and anhedonia in the 4 weeks prior to Screening.

Exclusion Criteria:

* Subjects who have received fluoxetine within 1 month prior to Baseline or any other antidepressant within 2 weeks prior to Baseline, or any unlicensed medication within 1 month before Screening
* Subjects who require psychotropic medication other than the study medication
* Subjects who started psychotherapy within 4 months prior to Screening
* Subjects who currently (i.e., in the month prior to Screening) meet DSM-IV criteria for bipolar syndrome or psychotic depression or severe somatoform or eating disorders
* Subjects who have a primary diagnosis of anxiety
* Subjects who regularly use sleeping medication more than 3 times per week
* Subjects who have major psychiatric or neurologic disorders other than MDD
* Subjects with depression secondary to stroke, cancer, or other severe medical illness
* Subjects who have a history of alcohol or substance dependence(within 1 year prior to Screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-11; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Björn Appelberg, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Department of Psychiatry
Locations (5):
- Finland (5):
  - Helsinki
  - Jyväskylä
  - Kuopio
  - Tampere
  - Turku